CLINICAL TRIAL: NCT00851058
Title: A Randomized Control Trial of the Effectiveness of of Group Motivational Counseling and an Emergency Department Experience in Reducing Risky Alcohol Use and Driving Behaviors.
Brief Title: Reducing Driving Offenses of Adolescent Drinkers
Acronym: ROAD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Ted Nirenberg PhD, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01AA15708-3; 5R01AA015708 (NIH)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Alcohol Consumption
Keywords: Behavioral research; Motivational counseling; Group Counseling; Motivational Interviewing; Vicarious Learning; Risky alcohol use; Recidivism; Motor Vehicles; Crime
MeSH Terms: conditions — Alcohol Drinking; Recidivism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Counseling (Experimental): Four session of group counseling and six hours of guided observation of the emergency and trauma services at a busy urban hospital
  Interventions: Behavioral: Brief group counseling
- Community Counseling (Active Comparator): Four session of group counseling and six hours of volunteering in a local not for profit community agency.
  Interventions: Behavioral: Community Counseling
- Prototypic Community Service (Placebo Comparator): Four hours of education about road safety and 16 hours volunteering at a local not for profit community service.
  Interventions: Behavioral: Prototypic community service

INTERVENTIONS:
Behavioral: Brief group counseling — Four group counseling sessions and six hours of direct observations of the emergency and trauma services in a busy urban hospital.
  Arms: Counseling
Behavioral: Community Counseling — Four session of group counseling and six hours of guided observation of the emergency and trauma services at a busy urban hospital
  Arms: Community Counseling
Behavioral: Prototypic community service — Two educational session on road safety and 16 hours of volunteering in a local not for profit community service.
  Arms: Prototypic Community Service
Behavioral: Prototypic community service — Four hours education about road safety and 16 hours volunteering at a local not for profit community service
  Arms: Prototypic Community Service

SUMMARY:
To determine the effectiveness of four group session of motivational counseling plus six hours of direct observations of the emergency department trauma services in comparison to four group session and six hours of community volunteering and also in comparison to four hours of education and 16 hours of community volunteering in reducing alcohol use and high risk driving behaviors and offenses among court referred 16-20 year old drivers.

ELIGIBILITY:
Age 16-20 years:

* Court referral for driving conviction and/or possession of alcohol
* Offense committed in Rhode Island
* Can speak English

Exclusion Criteria:

* Age over 20 years
* Not English speaking
* Not referred by courts

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 786 (Estimated)
Dates: Start 2007-05; Primary Completion 2010-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Recidivism for future criminal offenses | 12 months post intervention completion

SECONDARY OUTCOMES:
Alcohol use | 12 months post intervention completion

CONTACTS AND LOCATIONS:
Overall Officials: Ted D Nirenberg, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States